CLINICAL TRIAL: NCT03684109
Title: Pilot Study for Non-invasive Glioma Characterization Through Molecular Imaging
Brief Title: Non-invasive Glioma Characterization Through Molecular Imaging
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Macarena De La Fuente, MD, Assistance Professor, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20180606
Record Dates: First submitted 2018-09-21; First posted 2018-09-25 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Glioma; Brain Tumor; Primary Brain Tumor; Malignant Glioma; Malignant Primary Brain Tumor
Keywords: Non-invasive glioma characterization; Molecular Imaging; Isocitrate Dehydrogenase (IDH) Mutations; MRI-Based Sequencing
MeSH Terms: conditions — Glioma; Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- IDH-Mutant Glioma Patients (Experimental): Patients who have suspected or confirmed gliomas and are scheduled to undergo biopsy or resection of their brain tumors will receive a 3 Tesla (3T) Magnetic Resonance Imaging (MRI) scan of their brain.
  Interventions: Device: 3T MRI Scanner

INTERVENTIONS:
Device: 3T MRI Scanner — 3T MRI Scanner providing Mega-laser sequence for single-voxel Magnetic Resonance Spectroscopy (MRS) data for 2 hydroxyglutarate (2HG) quantitation.
  Other Names: 3 Tesla (3T) Magnetic Resonance Imaging Scanner

SUMMARY:
MRI-based sequences can provide non-invasive quantification of intratumoral 2-hydroxyglutarate (2HG) distribution and tumor cellularity in human gliomas and help guide the development of novel glioma therapies.

DETAILED DESCRIPTION:
This is a pilot study aiming at developing and optimizing MRI-based sequences to provide non-invasive quantification of intratumoral 2-hydroxyglutarate (2HG) distribution and tumor cellularity in human gliomas and help guide the development of novel glioma therapies.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 year old)
* Subjects with suspected or confirmed gliomas and who will have a medically indicated biopsy or resection of his/her brain lesion.

Exclusion Criteria:

* Adults unable to consent
* Individuals who are not yet adults (infants, children, teenagers)
* Pregnant women
* Patients unable to have MRI done

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-01-25 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
2HG Concentration via 3T MRI Scanner | Day 1
  2HG concentrations as measured via 3T MRI Scanner.
2HG Concentration from tissue samples | Day 1
  2HG concentrations as measured via patient's surgically excised tissue sample ex vivo by tissue based liquid chromatography-mass spectrometry (LC-MS)

CONTACTS AND LOCATIONS:
Overall Officials: Macarena De La Fuente, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No